CLINICAL TRIAL: NCT01505751
Title: The Association of G9a Protein and the Outcome of Patients With Cervical Cancer
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 100078-E
Record Dates: First submitted 2011-12-27; First posted 2012-01-09 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2015-07

CONDITIONS: Cervical Cancer
Keywords: Outcome of cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Residual pathology block after pathological exam

GROUPS / COHORTS (1):
- cervical cancer

SUMMARY:
G9a protein was approved to be highly associated with recurrence of breast cancer, gastric cancer, hepatocellular cancer, prostate cancer and lung cancer. Therefore, the aim of this study was to clarify the association and G9a protein and cervical cancer by analyzing the immunohistochemical staining of G9a protein to the histopathologic specimen of cervical cancer and clinical data.

ELIGIBILITY:
Inclusion Criteria:

* cases with cervical cancer

Ages: 20 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cervical cancer, and underwent primary treatment (surgery, radiotherapy or chemotherapy) in Far Eastern Memorial Hospital
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2012-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
determine whether G9a protein is a risk factor of overall survival of patients with cervical cancer | From the date of primary treatment until the date of death from any cause or the date of last follow-up, whichever came first, assessed up to 100 months

SECONDARY OUTCOMES:
determine whether G9a protein is a risk factor of progression-free survival of patients with cervical cancer | From the date of primary treatment until the date of first documented progression or last follow-up, whichever came first, assessed up to 100 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far-Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan